CLINICAL TRIAL: NCT01499394
Title: The Caris Biorepository Research Protocol
Brief Title: Caris Biorepository Research Protocol
Status: Recruiting | Type: Observational
Sponsor: Caris Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TCBIO-001-0710
Record Dates: First submitted 2011-12-16; First posted 2011-12-26 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Early Detection of Cancer; Minimal Residual Disease
Keywords: Caris Biorepository; MCED; Early Detection; MRD; Pan-Cancer
MeSH Terms: conditions — Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Currently plasma with an opportunity to collect other biospecimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Normal: Donor samples reflective of a "normal" non-disease state
- Newly Diagnosed Pan-Cancer Collection: Donor samples derived from treatment naïve patients with newly diagnosed solid tumors.
- Early Detection Collection: Donor samples reflective of a population at increased risk for developing cancer.
- Advanced Stage Cancer Collection: Donor samples derived from individuals with advanced stage cancer.
- Minimal Residual Disease Collection: Donor samples obtained from individuals with a history of malignancy who are currently free of active disease

SUMMARY:
The Biorepository for Caris Life Sciences is designed for the purpose of making quality biospecimens and associated clinical data available for research studies related to advancing precision medicine and improving care for patients.

The Caris Biorepository is a repository of prospectively collected biological specimens and associated clinical and demographic data gathered from multiple sources to be stored, used and shared for research. Caris Life Sciences will maintain the data and specimens and will control access to and use of the information and specimens by multiple individuals for multiple purposes which may evolve over time.

DETAILED DESCRIPTION:
The Caris Biorepository is an effort toward defining the future of medicine incorporating the discoveries of the genomic era by providing physicians, researchers and scientists access to quality human specimens and data aimed at improving human health and fighting disease. This will be accomplished through acquiring and sharing valuable biospecimen information and clinical outcomes in a collaborative, secure environment. The Caris Biorepository will bridge the gap and correlate human specimens with clinical and specimen data valuable to multiple and varying entities interested in advancing science with precision medicine by targeting disease treatments.

The objective of this project is to develop and implement a state-of-the-science Biorepository that ensures molecular integrity and clinical relevance of human biospecimens used in research and clinical medicine. The Caris Biorepository will also provide vital biospecimens and data to internal researchers and external research collaborators such as government, academia and industry collaborators for the use of drug development discoveries, clinically relevant research trials, publications and posters, and the implementation of future healthcare policies. This project may also impact characterization of trends in practice patterns and their relation to patient outcomes as well as the economic implications of differing evaluation, treatment and management paradigms.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Capacity to provide informed consent

Exclusion Criteria:

* Due to the complexity of state and federal requirements governing the participation of prisoners in research, prisoners-patients will not be approached for participation in the Caris Biorepository.
* Minor subjects will not be included in the Caris Biorepository, as it is possible biospecimens and data may be stored beyond the time limitations of assent and it may be impracticable to re-consent these subjects once they become adults.
* Individuals who lack the capacity to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers as well as those with a known disease state or condition
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2010-11; Primary Completion 2030-11 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
Develop biorepository that ensures molecular integrity and clinical relevance of quality human biospecimens and associated clinical data. | 35 years
  Retention of biospecimen samples with DNA
Implement release of specimens from biorepository for testing | 35 years
  Research for the purposes of cancer laboratory diagnostic tests.

SECONDARY OUTCOMES:
Laboratory testing | 35 years
  DNA and RNA microarray
Laboratory testing | 35 years
  Immunohistochemistry
Laboratory testing | 35 years
  Gene and protein expression, proteomics and matabolomics
Laboratory testing | 35 years
  Mutation analysis
Laboratory testing | 35 years
  Experiemental lab testing for development of new diagnostic technology
Laboratory testing | 35 years
  Microvesicle discovery, characterization and validation.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Oberley, MD, Principal Investigator — Caris Life Sciences
Locations (38):
- United States (38):
  - University of South Alabama, Mobile, Alabama
  - Southwest Medical Imaging, Scottsdale, Arizona
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - ObjectiveHealth - ARcare Center for Clinical Research, Little Rock, Arkansas
  - Lee Memorial Health System, Fort Myers, Florida
  - Cancer Care of North Florida, Lake City, Florida
  - Advent Health, Orlando, Florida
  - The University of South Florida, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Emory University, Atlanta, Georgia
  - Augusta University Research Institute, Augusta, Georgia
  - Cancer Center of Middle Georgia, Dublin, Georgia
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - CHRISTUS - St. Frances Cabrini Hospital, Alexandria, Louisiana
  - Tulane University, New Orleans, Louisiana
  - CHRISTUS - Highland Medical Center, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Jackson Oncology Associates, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - ObjectiveHealth - Premier Health Research, Sparta, New Jersey
  - CHRISTUS - St. Vincent Regional Cancer Center, Santa Fe, New Mexico
  - St. Lawrence Health System, Potsdam, New York
  - National Translational Research Group, Ridge, New York
  - Altru Health System, Grand Forks, North Dakota
  - NEO Urology Associates, Boardman, Ohio
  - Great Lakes Medical Research, Cleveland, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - Clinical Biotechnology Research Institute at RSFH, Charleston, South Carolina
  - Spartanburg Regional Health Services, Spartanburg, South Carolina
  - West Cancer Center, Germantown, Tennessee
  - ObjectiveHealth - Amarillo Premier Research, Amarillo, Texas
  - CHRISTUS - St. Michael's Health, Texarkana, Texas
  - CAMC Clinical Trials, Charleston, West Virginia
  - Mercy Health, Janesville, Wisconsin